CLINICAL TRIAL: NCT02018900
Title: The Effects of the Synbiotic Ecologic 825/scFOS on Intestinal Barrier Function
Brief Title: The Effects of the Synbiotic Ecologic 825/scFOS on Intestinal Barrier Function and Immune Modulation
Acronym: CRIB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-3-016
Record Dates: First submitted 2013-12-09; First posted 2013-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Volunteers
Keywords: Synbiotics; Intestinal permeability; Microbiota; Immune response

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Ecologic 825/scFOS (Experimental): Ecologic 825/scFOS
  Interventions: Dietary Supplement: Ecologic 825/scFOS

INTERVENTIONS:
Dietary Supplement: Ecologic 825/scFOS
  Arms: Ecologic 825/scFOS
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
In the present pilot study, the investigators will study the effects of a novel synbiotic, which is a mix of probiotics (Ecologic 825) in the presence of a prebiotic (short chain fructo-oligosaccharide (scFOS)), on mucosal integrity, overall microbiota changes along the gastrointestinal-tract and the mucosal immune response. The investigators hypothesize that the synbiotic Ecologic 825/scFOS will significantly affect the intestinal permeability and modulate the immune system in humans.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous self-admitted examination, no gastrointestinal complaints can be defined
* Age between 18 and 65 years
* Body Mass Index (BMI) between 20 and 30 kilogram/m2

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, head, ears, eyes, nose, throat (HEENT), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. - Use of medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing
* Administration of probiotic supplements, investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Use of antibiotics in the 90 days prior to the study
* Abdominal surgery interfering with gastrointestinal function, upon judgment of the principle investigator)
* Pregnancy, lactation
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* Smoking
* Blood donation within 3 months before or after the study period
* Self-admitted Human immunodeficiency virus-positive state
* History of any side effects towards intake of pro- or prebiotic supplements of any kind

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Sugar recovery in urine, as indicator of intestinal permeability | Baseline and after 2 weeks intervention

SECONDARY OUTCOMES:
Biomarkers of immune modulation; plasma levels of Tumor necrosis factor alpha , Interleukin-1 beta, Interleukin-6, Interleukin-8, Interleukin-17, Monocyte chemoattractant protein-1 and Macrophage inflammatory protein-1a | Baseline and after 2 weeks intervention
Relative abundance of commensal rat ileum bacterium (CRIB) by quantitative polymerase chain reaction (qPCR) | Baseline and after 2 weeks intervention
Barcoded pyrosequencing of 16S rRNA genes of the microbiota | Baseline and after 2 weeks intervention
Metatranscriptomics of the microbiota | Baseline and after 2 weeks intervention
10 item gastrointestinal symptom diary | Baseline and after 2 weeks intervention
Quantitative Insights Into Microbial Ecology (QIIME) of the microbiota | Baseline and after 2 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: A.A.M. Masclee, Professor, Principal Investigator — Department of Internal Medicine, Division of Gastroenterology-Hepatology
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] An R, Wilms E, Gerritsen J, Kim HK, Perez CS, Besseling-van der Vaart I, Jonkers DMAE, Rijkers GT, de Vos WM, Masclee AAM, Zoetendal EG, Troost FJ, Smidt H. Spatio-temporal dynamics of the human small intestinal microbiome and its response to a synbiotic. Gut Microbes. 2024 Jan-Dec;16(1):2350173. doi: 10.1080/19490976.2024.2350173. Epub 2024 May 13. PMID 38738780